CLINICAL TRIAL: NCT07050771
Title: Comprehensive Multimodal Prehabilitation Alone or in Combination With Planned Neoadjuvant Therapy in High-risk Patients Prior to Elective Major Cancer Surgery
Brief Title: Comprehensive Multimodal Prehabilitation Alone or With Neoadjuvant Therapy Before Major Cancer Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Nestor Esnaola, Professor of Surgery, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00039923
Record Dates: First submitted 2025-05-07; First posted 2025-07-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hepatopancreaticobiliary (HPB) Malignancy; Ovarian Cancer (OvCa); Kidney Cancers; Bladder Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive the pre-surgery CMMP only or CMMP with neoadjuvant therapy, based on their cancer characteristics and clinical needs. The CMMP consists of at least 3 weeks of therapy (nutritional supplements, exercise, and motivational interviewing). After surgery, 30-day morbidity-free survival will be determined and compared to historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMMP intervention (Experimental): Participants will receive the CMMP intervention, which includes motivational interviewing, nutritional prehabilitation (nutritional assessment/counseling and protein supplementation), inspiratory muscle training, and physical prehabilitation (aerobic and strength/resistance training) for at least 3 weeks prior to elective major cancer surgery.
  Interventions: Other: Comprehensive multimodal prehabilitation (CMMP)
- Planned neoadjuvant therapy/CMMP intervention (Experimental): Participants will receive the CMMP intervention (in conjunction with planned, off-protocol neoadjuvant therapy), which includes motivational interviewing, nutritional prehabilitation (nutritional assessment/counseling and protein supplementation), inspiratory muscle training, and physical prehabilitation (aerobic and strength/resistance training) for at least 3 weeks prior to elective major cancer surgery.
  Interventions: Other: Comprehensive multimodal prehabilitation (CMMP)

INTERVENTIONS:
Other: Comprehensive multimodal prehabilitation (CMMP) — Components of the CMMP intervention (which will be administered for at least 3 weeks from study registration to the Preoperative Reassessment) will include: 1) Motivational interviewing: 2 sessions, 10-15 minutes each. 2) Nutritional prehabilitation (a supplement containing 18-22g high quality protein consumed 2 times/day, 7 days/week). 3) Inspiratory muscle training using a hand-held inspiratory muscle device, 5 minutes of respiratory muscle training twice/day, 5 days per week. 4) Physical prehabilitation a) aerobic exercise (20 minutes of moderate-intensity exercise at least 3 days/week) and b) strength resistance training using resistance bands (3 sets of 10 repetitions at moderate intensity at least 3 days/week).

SUMMARY:
In this 2-arm, non-randomized, phase II trial, the investigators will evaluate the efficacy and safety of comprehensive multimodal prehabilitation (CMMP) alone or in combination with planned neoadjuvant (NAT) in pre-frail/frail patients with probable/proven pancreaticobiliary, ovarian, kidney, or bladder cancer prior to elective major cancer surgery (EMCS).

DETAILED DESCRIPTION:
This is a 2-arm, non-randomized, phase II trial evaluating the efficacy and safety of comprehensive multimodal prehabilitation (CMMP) alone or in combination with planned/off-protocol neoadjuvant therapy (NAT) in high-risk (pre-frail/frail) patients with probable/proven pancreaticobiliary, ovarian, renal, or bladder cancer prior to elective major cancer surgery (EMCS, including pancreatectomy [N=38 in each study arm], cytoreduction [N=12 in each study arm], radical nephrectomy [N=12 in each study arm], or total cystectomy [N=12 in each study arm]; respectively and accounting for a potential 20% dropout rate). The two study arms are independent; within arm (i.e., across cancer and/or procedure types) and between arm comparison will not be performed. The CMMP intervention combines motivational interviewing (MI) with nutritional prehabilitation, inspiratory muscle training, and physical prehabilitation (aerobic exercises and strength/resistance training). Approximately 74 high-risk, male or female patients, 18 years of age or older, will be enrolled in Arm 1 (CMMP alone) and 74 similar patients will be enrolled in Arm 2 (CMMP & planned NAT).

The primary endpoints are postoperative morbidity-free survival and safety after CMMP. The secondary endpoints are preoperative functional status/fitness; completion of planned preoperative therapy (in Arm 2 only); preoperative/postoperative health-related quality-of -life (HRQOL); and receipt of intended (adjuvant) oncologic therapy (RIOT). Additional secondary endpoints will include postoperative morbidity/healthcare utilization and 2-year overall survival (OS) and disease-free survival (DFS; in patients with proven [histologically confirmed] cancer) after CMMP. The tertiary endpoints are nutritional status and body composition after CMMP.

Exploratory analyses using baseline/pre-CMMP and post-CMMP peripheral blood samples, as well as baseline/pre-CMMP (clinical diagnostic biopsy) and post-CMMP (EMCS specimen) tumor samples will include (but not be limited to) correlates of response to CMMP including as peripheral immune modulation, as well as (in patients with proven cancer) changes to the tumor microenvironment (TME: vasculature, hypoxia, and immune cell infiltration) and pathologic response (in Arm 1 patients who did not receive NAT prior to study entry).

Patients in Arm 1 (CMMP alone) will receive (at least 3) weekly cycles of CMMP between study registration and Preoperative Reassessment. Patients in Arm 2 (CMMP & planned NAT) will receive (at least 3) weekly cycles of CMMP during receipt of planned/off-protocol NAT between study registration and Preoperative Reassessment. Patients will be provided with ready access to videos explaining the subcomponents of the CMMP intervention. Throughout the CMMP intervention, weekly automated assessments of adherence to the CMMP intervention and assessments for AEs/SAEs will be conducted electronically (via text/email using a text-enabled Research Electronic Data Capture [REDCap] database/system) and/or by study staff (in-person or by email/telephone).

At the Preoperative Reassessment, impact of the CMMP intervention on relevant intermediate endpoints will be evaluated, including, nutritional status, body composition (muscle mass), respiratory muscle function, muscular (grip) strength, functional capacity, functional status/fitness, HRQOL, and ECOG performance status.

After the Preoperative Reassessment, patients will proceed to planned/off protocol EMCS < 67 days after start of last cycle of CMMP. Patients who undergo EMCS and meet eligibility criteria at Second Registration will continue in the study and complete a series postoperative assessments, including assessments of postoperative mortality/morbidity, healthcare utilization, and HRQOL through postoperative day 90, as well as vital and (in patients with proven cancer) disease status assessments up to 2 years after First Registration.

Preoperative and postoperative peripheral blood and tumor tissue samples will be collected and used to conduct correlative studies exploring potential mechanism(s) of oncologic benefit of CMMP, including but to limited to changes in the peripheral immune milieu and (in patients with proven cancer) TME. Collection of blood specimens (PBMC, plasma, serum) will be performed at baseline (after First Registration) and at the Preoperative Reassessment; these specimens will be compared to assess peripheral immune modulation after CMMP. In patients with proven cancer, tumor tissue (in the form of slides) obtained as part of the patient's standard care (i.e., diagnostic biopsy) will be collected after First Registration and used to assess the pretreatment (baseline). Tumor tissue will also be collected at the time of EMCS (surgical resection specimen); these specimens will be compared to assess for changes in TME after the CMMP (and in patients in Arm 1 who did not received NAT prior to First Registration, as pathologic response to CMMP [alone]).

The investigators hypothesize that the CMMP intervention will be feasible and safe; improve preoperative nutritional status, muscle mass, and functional status/fitness; improve postoperative morbidity-free survival; improve perioperative HRQO; results in high rates of receipt of NAT and RIOT; and reduce postoperative PPCs and health care utilization. The investigators hypothesize that the CMMP intervention will result in peripheral immune mobilization and activation. In patients with proven cancer, the investigators further hypothesize that it will also result in improved tumor vasculature, reduced tumor hypoxia, and improved immune cell infiltration; and (even when used without NAT) potentially result in a pathologic response.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for entry into the study (First Registration) only if ALL of the following criteria apply. No exceptions or waivers will be granted for patients who do not meet the eligibility criteria.

* Signed informed consent form.
* Age ≥18 years at time of signing informed consent form.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 per the treating cancer surgeon (Arm 1, Neoadjuvant therapy) or per both the treating cancer surgeon and the medical and/or radiation oncologists (Arm 2, no neoadjuvant therapy).
* Pre-frail or frail (based on the Fried Frailty Phenotype
* Probable or proven (histologically confirmed) pancreaticobiliary/periampullary (i.e., pancreatic cancer, cholangiocarcinoma, duodenal cancer, or ampullary cancer), ovarian cancer, kidney cancer, or bladder cancer based on central pathological review at Houston Methodist Hospital.
* Clinically non-metastatic (stage I-III) or metastatic (IV) disease.
* Technically resectable disease (no significant vascular, neural, or bony involvement and potential to safely achieve R0 resection) and potentially medically fit for EMCS per the treating cancer surgeon (surgical oncologist/HBP surgeon, gynecologic oncologist, or urologic oncologist).
* Tentatively scheduled to undergo elective pancreatectomy (open or minimally invasive pancreaticoduodenectomy or open distal pancreatectomy) for pancreaticobiliary/periampullary cancer, elective surgical cytoreduction for ovarian cancer, elective open radical nephrectomy for kidney cancer, or elective (open or minimally invasive) total cystectomy for bladder cancer by one of the study MPI or Co-Is > 28 days after trial registration.
* Neoadjuvant therapy group only: Completed planned NAT (if any) at least 2 weeks prior to Study Registration.
* No neoadjuvant therapy group only: Medically fit and planned to receive NAT per the treating medical and/or radiation oncologist.
* Ability to comply with the CMMP intervention and study assessments as per protocol, in the MPI's judgment.
* Willing and able to consume a lactose-free, whey protein supplement (if not allergic to milk protein/soy and no history of galactosemia), marine protein supplement (if not allergic to marine protein/shellfish), or pea protein supplement (if not allergic to pea protein).
* Willing to provide tissue and blood specimens as per protocol.
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
* Access to a smart phone (personally or via caretaker who resides with the patient).
* Understands, speaks, and reads English.

Exclusion Criteria:

Patients are NOT eligible for entry into the study (First Registration) only ANY of the following criteria apply. No exceptions or waivers will be granted for patients who do not meet the eligibility criteria.

* Difficulty or inability to hear and/or understand loud speech and sounds.
* Unable to eat by mouth (e.g., tube feed dependent, on total parenteral nutrition, etc.)
* Oxygen dependent (or rest and/or with exertion).
* Significant cardiovascular disease (such as New York Heart Association (NYHA) Functional Classification III or IV, unstable angina, unstable arrhythmia, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of trial treatment.
* Dependence on mobility device for ambulation other than a cane (e.g., crutches, walker, wheelchair).
* Active brain metastasis or leptomeningeal disease.
* Active bone metastasis and/or recent bone fracture.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). NOTE: Patients with indwelling catheters (e.g., PleurX) are allowed
* Planned receipt of investigational therapy/treatment (other than the protocol-mandated CMMP intervention) during the trial treatment.
* Major procedure/surgery within 12 weeks prior to initiation of trial treatment that would prevent the patient from complying with the CMMP intervention and study assessments as per protocol, in the MPI's judgment.
* Active physical/mental condition or personal/social circumstance that would prevent the patient from complying with the CMMP intervention and study assessments as per protocol, in the MPI's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of morbidity-free survival | At 30 days postoperatively
  Percentage of patients alive without any postoperative complications (as defined by the American College of Surgeons National Surgical Quality Improvement Program {ACS NSQIP]) in each study arm.
Rates of adverse events and serious adverse events | From study enrollment to the time of planned, off-protocol, preoperative re-evaluation by the participant's primary cancer surgeon (approximately 1 month after enrollment in Arm 1 and 2-3 months after enrollment in Arm 2 ).
  Percentage of patients with adverse events and serious adverse events (AEs/SAEs; as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0) during receipt of CMMP in each study arm.

SECONDARY OUTCOMES:
Rate of improvement in preoperative functional status/fitness | At the time of planned, off-protocol, preoperative re-evaluation by the participant's primary cancer surgeon (approximately 1 month after enrollment in Arm 1 and 2-3 months after enrollment in Arm 2).
  Percentage of patients in each study arm with improvement (compared to baseline) in > 2 of the following measures of functional status/fitness at the Preoperative Reassessment: change in maximal inspiratory pressure (MIP) by > 19 cmH2O, change in grip strength by > 5 kgs; and/or change in gait speed by > 0.1m/s
Rate of completion of planned preoperative therapy | At the time of planned, off-protocol, preoperative re-evaluation by the participant's primary cancer surgeon (approximately 1 month after enrollment in Arm 1 and 2-3 months after enrollment in Arm 2).
  Percentage of patients in Arm 2 who completed their planned preoperative therapy
Health-related quality of life (HRQOL) | At the time of planned, off-protocol, preoperative re-evaluation by the participant's primary cancer surgeon (approximately 1 month after enrollment in Arm 1 and 2-3 months after enrollment in Arm 2) and at 30, 60, and 90 days postoperatively.
  Change in HRQOL (based on the Short Form [SF]-12; compared to baseline) in each study arm. More specifically, changes in the Mental Health Component (MCS; range 3.2-77.9) and the Physical Health Component (PCS; range 9.9-76) will be analyzed (higher scores indicate better HRQOL with respect to that component).
Postoperative rate of receipt of intended oncologic therapy (RIOT) | At 30, 60, and 90 days postoperatively
  Percentage of patients who received planned (intended) oncologic therapy after EMCS in each study arm
Rate of postoperative pulmonary complications (PPCs) | At 30 days postoperatively
  Percentage of patients with PPCs (ventilator > 48 hours, unplanned intubation, and/or pneumonia; as defined by ACS NSQIP) in each study arm
Rate of postoperative discharge to home | At the time of hospital discharge (approximately 7 days postoperatively)
  Percentage of patients discharged to home after EMCS in each study arm
Rate of hospital readmission | At 30, 60, and 90 days postoperatively
  Percentage of patients readmitted to hospital (as defined by ACS NSQIP) after EMCS in each study arm
Postoperative length of stay | At the time of hospital discharge (approximately 7 days postoperatively)
  Number of days from date of EMCS to date of hospital discharge in each study arm
Overall survival (OS) | 2 years after EMCS
  OS in each study arm
Disease-free survival (DFS) | 2 years after EMCS
  DSF (in patients with proven cancer at EMCS) in each study arm

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: SAP, ICF
Time Frame: After publication of primary study outcomes
Access Criteria: Other investigators; via an emailed and approved proposal that describes planned analyses and a signed data sharing agreement.